CLINICAL TRIAL: NCT07061366
Title: The Use of the Bambi-Belt in Exteremly Preterm Infants: an Implementation Study
Acronym: BB-EP
Status: Recruiting | Type: Observational
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Hendrik Niemarkt, Principal investigator, Maxima Medical Center
Other Study IDs: N25.024
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Preterm; Monitoring
Keywords: wireless; monitoring; heart rate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extremely preterm infants

SUMMARY:
This observational, non-interventional cohort study evaluates the clinical use of the Bambi Belt-a CE-certified, wireless device for non-invasive heart rate and respiration monitoring-in extremely preterm infants (<26 weeks gestation). 15 infants with intact skin and age <24 hours will be monitored using the Bambi Belt during the first ten days of life. Primary outcomes include ease of use (application, signal stability), skin tolerance, and user experience (nurses and parents). Standard care remains unchanged. Data will be collected via clinical records and evaluation forms.

DETAILED DESCRIPTION:
The Bambi Belt is a CE-certified, wireless monitoring device designed for continuous, non-invasive measurement of heart rate and respiration in neonates. Developed and validated in our center, it offers several advantages over traditional adhesive electrodes, including reduced skin irritation, improved comfort during kangaroo care, and easier handling of the infant. These features are particularly relevant for extremely preterm infants (<26 weeks gestation), whose skin is highly vulnerable and for whom standard electrodes often pose clinical challenges.

Following a successful implementation phase in the general neonatal population, this study aims to evaluate the use of the Bambi Belt specifically in extremely preterm infants. Because of the low prevalence of this group, targeted implementation has not yet occurred. This observational cohort study will include 15 infants who meet the following inclusion criteria: gestational age <26 weeks, postnatal age <24 hours, and intact skin.

The Bambi Belt will be used as the standard method for heart rate and respiration monitoring during the first ten days of life. All other aspects of care remain unchanged. Outcomes will focus on:

Ease of use: including the ease of application, signal stability, and frequency of repositioning.

Skin tolerance: assessment of any skin reactions that necessitate switching back to conventional electrodes.

User experience: qualitative feedback from nurses and parents, collected via brief evaluation forms.

Clinical data will be obtained from the hospital's electronic patient record system (EPD/DWH). All data will be coded and processed according to GDPR and institutional guidelines. Parents will provide informed consent, including optional consent for anonymous data sharing with the device manufacturer (Bambi Medical).

This study is classified as non-WMO research, based on the minimal risk to the patient and the fact that the device is CE-marked and used within its intended purpose. The prior implementation phase has already been reviewed and approved as non-WMO by our local ethics review committee

ELIGIBILITY:
Inclusion Criteria: Preterm born <26 weeks; first week of life -

Exclusion Criteria: skin integrity problems prior to study, palliative care.

-

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely preterm infants in NICU
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Ease of use | As long as belt is worn (10 days)
  ease of application according to score of nurse.
Skin integrity | as long as belt is worn (10 days)
  any skin reactions that necessitate a switch back to conventional electrodes
User experience | From belt is worn till month after
  feedback from nurses and parents, collected through brief evaluation forms
Signal stability | during 10 days (study period wearing belt)
  Precentage of time were reliable respiratory and heart rate signal is collected

CONTACTS AND LOCATIONS:
Locations (1):
- Maxima Medical Centre, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scholten AWJ, Zhan Z, Niemarkt HJ, Vervoorn M, van Leuteren RW, de Jongh FH, van Kaam AH, Heuvel ERVD, Hutten GJ. Cardiorespiratory monitoring with a wireless and nonadhesive belt measuring diaphragm activity in preterm and term infants: A multicenter non-inferiority study. Pediatr Pulmonol. 2023 Dec;58(12):3574-3581. doi: 10.1002/ppul.26695. Epub 2023 Oct 5. PMID 37795597
- [Background] Lorente Flores CM, Zhan Z, Scholten AWJ, Hutten GJ, Vervoorn M, Niemarkt HJ. The Effects of a New Wireless Non-Adhesive Cardiorespiratory Monitoring Device on the Skin Conditions of Preterm Infants. Sensors (Basel). 2024 Feb 16;24(4):1258. doi: 10.3390/s24041258. PMID 38400415